CLINICAL TRIAL: NCT04358874
Title: Maximizing Acute Kidney Injury End-point Intervention Post-Discharge (MAKE-IT) Study
Acronym: MAKE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Vanderbilt University Medical Center (Other); University of Kentucky (Other)
Responsible Party: Principal Investigator, Orlando M. Gutierrez, MD, MMSc, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-161201002
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Medication Reconciliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active follow-up (Experimental): Participants randomized to the active follow-up arm will have follow-up visits in the AKI follow-up clinic every 4 weeks after discharge for a total of 90 days after discharge
  Interventions: Other: Medication reconciliation; Other: Blood Pressure Management
- Usual follow-up (Active Comparator): Participants randomized to the usual follow-up arm will be called at home 4 weeks after the baseline visit to collect information on primary and secondary outcomes.
  Interventions: Other: Medication reconciliation; Other: Blood Pressure Management

INTERVENTIONS:
Other: Medication reconciliation — Medicines currently being taken will be reviewed and compared to the medicines that were prescribed at discharge.
Other: Blood Pressure Management — Blood pressure will be checked at follow-up visits and medicines will be adjusted if blood pressure is above target range (>160/100)

SUMMARY:
This purpose of this pilot and feasibility study is to determine whether attending an acute kidney injury (AKI) clinic after discharge from the hospital impacts prescription medicine use, blood pressure and recovery of kidney function as compared to usual care.

DETAILED DESCRIPTION:
Participants with moderate to severe acute kidney injury (AKI) who are discharged from participating centers (the University of Alabama at Birmingham Hospital, Vanderbilt University Medical Center, University of Kentucky) will be randomized to coming to a dedicated AKI clinic at one of the three recruitment centers for up to four visits over 3 months or usual care. At the visits to the AKI follow-up clinics, medicine reconciliation will be done, blood pressure will be measured, information on hospitalizations and other adverse events will be taken and blood and urine samples will be collected to check kidney function and store samples to measure biomarkers of AKI. Participants randomized to usual care will be contacted by telephone to review medications currently being taken and to collect information on hospitalizations and other adverse events. The primary outcome measures will be include both process of care and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years and older
* Patients who have developed moderate to severe AKI in the hospital, defined as:

  1. At least a doubling of peak creatinine from baseline or receipt of dialysis while in the hospital
  2. AKI of any degree in individuals with an estimated glomerular filtration (eGFR) rate < 60 ml/min/1.73m2 at baseline
  3. AKI of any degree whose discharge creatinine does not return to within 50% of baseline.
* Able to provide signed informed consent

Exclusion Criteria:

* Patients with a history of kidney transplant
* Patients who, in the opinion of the investigator, are not suitable to participate in the study
* Unable to obtain written informed consent
* prisoners or pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Number of incorrectly prescribed medicines | 90 days
  The number of incorrectly dosed or prescribed medications that are detected or changed
Proportion of individuals restarting RAAS inhibitors | 90 days
  Proportion of patients with a class I indication for renin-angiotensin-aldosterone (RAAS) inhibitors who have appropriately re-started RAAS inhibitors within 3 months of discharge.
Blood pressure control | 90 days
  Systolic and diastolic blood pressure obtained by automatic blood pressure cuff in the clinic.
Recovery of kidney function | 90 days
  Proportion of individuals who have recovered from AKI, defined as a serum creatinine within 10% of baseline by 3 months

SECONDARY OUTCOMES:
Major adverse kidney outcomes | 90 days
  Defined as a composite of death, need for new dialysis, rehospitalization for AKI, recurrent AKI, or a persistent increase in baseline serum creatinine of ≥ 50%.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - University of Kentucky, Lexington, Kentucky
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No